CLINICAL TRIAL: NCT05085496
Title: Phase I Trial of Radiotherapy in Combination With Atezolizumab in Borderline Resectable and Unresectable Cutaneous Squamous Cell Carcinoma(cSCC)
Brief Title: Radiotherapy in Combination With Atezolizumab in Locally Advanced Borderline Resectable or Unresectable Cutaneous SCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: Genentech, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21285; NCI-2021-09849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21285 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Skin Squamous Cell Carcinoma; Resectable Skin Squamous Cell Carcinoma; Unresectable Skin Squamous Cell Carcinoma
MeSH Terms: interventions — atezolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SBRT, atezolizumab) (Experimental): Patients undergo SBRT on days 1, 3, 5, 7, and 9 of cycle 1. Beginning 1-2 days after SBRT, patients also receive atezolizumab IV on day 1. Treatment repeats every 3 weeks for 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial tests the safety and side effects radiotherapy in combination with atezolizumab in treating patients with cutaneous squamous cell cancer that has spread to nearby tissue or lymph nodes (locally advanced) and can be removed from surgery (resectable) or cannot be remove by surgery (unresectable). Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving radiotherapy in combination with atezolizumab may help improve outcomes for remission (cancer that is under control) than taking either treatment separately.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety profile of combination of atezolizumab + radiation therapy (RT) in borderline resectable or unresectable cutaneous squamous cell carcinoma (cSCC).

SECONDARY OBJECTIVES:

I. Determine pathologic response after neoadjuvant atezolizumab + RT. II. Determine clinical response (via imaging and clinical exam) postoperatively (if surgically resectable) or at post-treatment biopsy (if not surgically resectable), and 3 months following the completion of surgery or RT (if not surgically resectable).

III. Define the toxicity profile associated with the treatment protocol. IV. Assess short-term quality-of-life associated with the treatment protocol.

EXPLORATORY OBJECTIVES:

I. To compare immune checkpoint molecule (e.g. PD1, PD-L1, TIM3, TIGIT, etc.) expression intensity within tumor cells and immune cells in the tumor microenvironment, as well as immune cell subset infiltration patterns including T cells before and after atezolizumab + stereotactic body radiation therapy (SBRT) by multiplex immunohistochemistry (or immunofluorescence).

II. To evaluate the impact of tumor molecular features on immune response and treatment outcome using next generation targeted deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) sequencing of pre-treatment tumor tissue.

III. To compare changes in circulating immune cell subsets in peripheral blood by RNA-based T-cell receptor (TCR)-sequencing and immunophenotyping by flow cytometry (or immunophenotyping by single-cell RNA sequencing), and correlate changes with response, clinical outcomes, and toxicity.

IV. To evaluate circulating tumor DNA (ctDNA) levels before start of treatment and immediately prior to surgery/repeat biopsy.

OUTLINE:

Patients undergo SBRT on days 1, 3, 5, 7, and 9 of cycle 1. Beginning 1-2 days after SBRT, patients also receive atezolizumab intravenously (IV) on day 1. Treatment repeats every 3 weeks for 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up every 12 weeks for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced borderline resectable or unresectable cSCC and oligometastatic (1-3 sites of metastatic disease) cSCC receiving therapy to the primary
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm with computed tomography (CT) scan or > 10 mm with calipers by clinical exam by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Written informed consent and any locally-required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States of America [USA], European Union [EU] Data Privacy Directive in the EU) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
* Age >= 18 years at time of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy >= 24 weeks
* Body weight > 30 kg
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (>= 1000 per mm^3)
* Platelet count >= 75 x 10^9/L (>= 75,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum albumin 25 g/L (2.5 g/dL)
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 3 months
* Patients with active interstitial lung disease (ILD)/pneumonitis or with a history of ILD/pneumonitis requiring steroids
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any previous treatment with a PD1 or PD-L1 inhibitor, including atezolizumab, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 30 days prior to the first dose of study drug for patients who have received prior tyrosine kinase inhibitors (TKIs) [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C. (If sufficient wash-out time has not occurred due to the schedule or pharmacokinetics (PK) properties of an agent, a longer wash-out period may be required.)
* Patients with corrected QT (QTc) interval > 470 msec during screening
* Current or prior use of immunosuppressive medication within 14 days (use 28 days if combining atezolizumab with a novel agent) before the first dose of atezolizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent

    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy that is not part of standard National Comprehensive Cancer Network (NCCN) indicated head and neck squamous cell carcinoma (HNSCC) adjuvant concurrent chemoradiotherapy (CRT). Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* History of allogenic organ or bone marrow transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, idiopathic pulmonary fibrosis, organizing pneumonia, uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently), uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium ULN), uncontrolled tumor-related pain, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 3 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive human immunodeficiency virus [HIV] 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving atezolizumab and up to 5 months after the last dose of atezolizumab
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 5 months after the last dose of atezolizumab monotherapy. Patient must have a negative serum pregnancy test within 72 hours of study entry
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Prior randomization or treatment in a previous atezolizumab clinical study
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 3 weeks
Incidence of adverse events | Up to 90 days
  Toxicity will be assessed by Common Terminology Criteria for Adverse Events version 5 criteria.

SECONDARY OUTCOMES:
Treatment response rate | After completion of cycle 3 (each cycle is 21 days)
  Will be calculated as the ratio of the number of patients who demonstrated a complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) divided by the number of patients evaluable for response.
Overall survival (OS) | From the date of diagnosis to the date of death, assessed up to 24 months
  Will be examined using the Kaplan-Meier method. Median OS and corresponding two-sided 95% confidence intervals will be computed.
Progression free survival (PFS) | From the date of diagnosis to the date of progression, assessed up to 24 months
  Will be examined using the Kaplan-Meier method. Median PFS and corresponding two-sided 95% confidence intervals will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States